CLINICAL TRIAL: NCT06161909
Title: Postoperative Adjuvant Immune Maintenance Therapy for High Recurrence Risk Esophageal Squamous Cell Carcinoma After Radical Resection: a Multicenter Randomized Controlled Clinical Trial
Brief Title: Postoperative Immune Maintenance Therapy for Esophageal Squamous Cell Carcinoma After Radical Resection
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: POSLS-union02
Record Dates: First submitted 2023-11-22; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-10

CONDITIONS: Esophageal Squamous Cell Carcinoma Thoracic Stage II; Esophageal Squamous Cell Carcinoma Thoracic Stage III; Esophageal Squamous Cell Carcinoma Thoracic Stage IV
Keywords: Esophageal cancer; Surgery; Immunotherapy; Prognosis
MeSH Terms: conditions — Esophageal Neoplasms | interventions — sintilimab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Postoperative adjuvant sintilimab 200mg fixed dose Q3W, immunotherapy will be administered for a total of 1 year.
  Interventions: Drug: sintilimab
- Group B (No Intervention): Close observation.

INTERVENTIONS:
Drug: sintilimab — 200mg fixed dose Q3W,1 year
  Arms: Group A

SUMMARY:
Esophageal cancer (EC) is one of the most common malignant tumors of the digestive tract in human beings. Most cases of EC are initially diagnosed in an advanced stage of the disease. Considering the lack of effective adjuvant therapies after surgery for locally advanced esophageal squamous carcinoma. And with the encouraging preliminary results of PD-1 inhibitors in advanced esophageal squamous cell carcinoma (ESCC), postoperative adjuvant immunotherapy for esophageal squamous carcinoma seems to be feasible. The main objective of this study was the efficacy of postoperative adjuvant therapy with sintilimab in patients with ESCC radically resected after neoadjuvant chemoimmunotherapy.

DETAILED DESCRIPTION:
sophageal cancer (EC) is one of the most common malignant tumors of the digestive tract in human beings. Most cases of EC are initially diagnosed in an advanced stage of the disease. Considering the lack of effective adjuvant therapies after surgery for locally advanced esophageal squamous carcinoma. And with the encouraging preliminary results of PD-1 inhibitors in advanced esophageal squamous cell carcinoma (ESCC), postoperative adjuvant immunotherapy for esophageal squamous carcinoma seems to be feasible. The main objective of this study was the efficacy of postoperative adjuvant therapy with sintilimab in patients with ESCC radically resected after neoadjuvant chemoimmunotherapy.

All participants who meet the inclusion criteria will be enrolled after signing the informed consent form. A total of 400 patients are to be recruited for the study. 400 subjects were randomly assigned to the two treatment groups. Group A: Postoperative adjuvant sintilimab 200mg fixed dose Q3W, immunotherapy will be administered for a total of 1 year. Group B: Close observation. The primary endpoint is disease-free survival (DFS). The secondary endpoints are postoperative overall survival (OS); 1, 2, and 3-year postoperative OS rates; recurrent metastasis pattern (local recurrence or distant metastasis).

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to the implementation of any trial-related processes;
2. Male or female, ≥18 years of age or ≤75 years of age;
3. Pathologically confirmed ESCC in the thoracic segment;
4. Received 2-4 cycles of neoadjuvant chemoimmunotherapy and assessed by imaging as CR or PR (clinical staging of cT1b-T2,N+ or cT3-T4a,ANY N) (8th edition UICC/AJCC TNM staging);
5. Underwent radical surgery, and had negative surgical margins confirmed pathologically after surgery (R0), defined as the absence of squamous carcinoma cells from the proximal, distal, or peripheral resection borders of esophageal carcinoma;
6. Postoperative pathological assessment of non-pCR, and residual tumor in the primary tumor focus or regional lymph nodes.

Exclusion Criteria:

1. Patients with an untreated diagnosis of another malignancy within 5 years prior to the first dose (excluding radically treated basal cell carcinoma of the skin, squamous epithelial carcinoma of the skin, and/or carcinoma in situ that has undergone radical resection);
2. Serious surgical complications after resection of esophageal cancer with reference to Clavien-Dindo classification > 3;
3. Individuals with a history of allergy or hypersensitivity to components of the study drug or severe hypersensitivity to any monoclonal antibody;
4. All toxicities (other than nephropathy, neuropathy, hearing loss, alopecia, and fatigue) attributable to prior antitumor therapy (preoperative induction therapy) must have recovered to baseline levels or Grade 1 (CTCAE Version 5.0) prior to administration of study drug;
5. Received systemic therapy with a proprietary medicine with an antitumor indication or an immunomodulatory drug (including thymidine, interferon, interleukin, except for local use to control pleural fluid) within 2 weeks prior to the first dose;
6. Women who are pregnant or breastfeeding;
7. Presence of any serious or uncontrollable systemic disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-01-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
disease-free survival (DFS) | 2 years
  disease-free survival (the time from the date of randomization to the first date of disease recurrence or death, whichever occurred first, before subsequent anticancer therapy).DFS for 400 participants.

SECONDARY OUTCOMES:
postoperative overall survival (OS) | 2 years
  The postoperative overall survival (OS) was defined as the time from primary tumor resection (surgical date) to last follow-up or death.OS for 400 participants.
1, 2, and 3-year postoperative OS | 1, 2, and 3-year
  1, 2, and 3-year postoperative OS for 400 participants.
recurrent metastasis pattern | two-year period
  recurrent metastasis pattern (local recurrence or distant metastasis) for 400 participants.

CONTACTS AND LOCATIONS:
Overall Officials: Maohui Chen, Study Chair — Fujian Medical University Union Hospital
Locations (1):
- Fujian, Fujian, China